CLINICAL TRIAL: NCT01381263
Title: Development, Evaluation and Cost Effectiveness of a Treatment Program With a Behavioural Medicine Approach for Adolescents With Persistent Pain.
Brief Title: Behavioral Medicine Treatment for Adolescents in Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: The Swedish Research Council (Other Government); Uppsala County Council, Sweden (Other Government)
Responsible Party: Anne Söderlund, professor, University of Uppsala Department of Neuroscience
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dnr 2010/047
Record Dates: First submitted 2010-12-20; First posted 2011-06-27 (Estimated); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioural medicine (Experimental)
  Interventions: Behavioral: Behavioural medicine treatment
- Standard treatment (Active Comparator): Standard treatment includes muscle strengthening, stretching, posture training, training of relaxation techniques and information about pain according to the best empirical praxis
  Interventions: Other: Standard treatment

INTERVENTIONS:
Behavioral: Behavioural medicine treatment — The behavioural medicine treatment program will include muscle strengthening, stretching, posture training, training of relaxation techniques and information about pain according to the best empirical praxis and age appropriate interventions aimed to address the emotional and behavioural processes of pain.
  Arms: Behavioural medicine
Other: Standard treatment — Standard treatment includes muscle strengthening, stretching, posture training, training of relaxation techniques and information about pain according to the best empirical praxis
  Arms: Standard treatment

SUMMARY:
Recurrent pain, such as headache, stomach pain and musculoskeletal pain is common in children and adolescents. Children and adolescents are reported to have restrictions in daily life activities, social contacts, and school attendance, and to have poorer academic skills and as well as an increased utilization of heath care services due to pain problems. The treatment approaches available today for teenagers with pain are often biological/physiological and little evidence for their effectiveness has been shown. It is urgent to try new interventions for pain problems in early ages in order to prevent disability, development of maladaptive coping strategies and to avoid negative impact on daily activities.

The optimal treatment regime for paediatric pain patients has been suggested to be cognitive behavioural approach integrated with physical therapy The aim of this project is to develop and evaluate in a randomized controlled trial a treatment program with a behavioural medicine approach (suitable to use in primary care or school based health care context) compared with standard treatment for adolescents with persistent pain problems. The aim is also to compare short and long-term costs for patients and for the health care system related to the two interventions, in order to determine strategies for future cost-effective care of children and adolescents experiencing recurrent pain.

DETAILED DESCRIPTION:
Chronic or recurrent pain symptoms are widely studied and generally regarded as an important public health concern in adults. The prevalence of pain symptoms are reported to be as high as 25-30 % in children and adolescents. Children and adolescents are reported to have restrictions in daily life activities, social contacts, and school attendance, and to have poorer academic skills and as well as an increased utilization of heath care services due to pain problems. These patients suffer from a wide variety of problems, for example sports injuries, persistent postoperative pain, musculoskeletal pains, headaches or multiple recurrent pain problems. The treatments given today to adolescents are dealing with symptoms in a physical manner.

In this study participants will be recruited among adolescents referred to paediatric physiotherapy. The participants will be randomly allocated to either physiotherapy including standard treatment or a behavioural medicine treatment program. Standard treatment includes muscle strengthening, stretching, posture training, training of relaxation techniques and information about pain according to the best empirical praxis.

The behavioural medicine treatment program will include the same components as the standard treatment with the addition of age appropriate interventions aimed to address the emotional and behavioural processes of pain. The treatment is based on earlier intervention programs and includes the following phases;

* Individual functional behavioural analysis The adolescents lists specific important and frequent activities and situations they have problems to master due to pain and target activities are then chosen. Individual capabilities (both physical and psychological), behavioural responses, and their short and long-term consequences are identified. Parental responses and their impact on adolescent's pain behaviours are noted. Target activity related treatment goals as well goals for engagement in the treatment are defined from the individual functional behavioural analysis.
* Basic skill acquisition Physical abilities and cognitive skills required for improvement of behaviour in target activities are trained. For example to meet the problem of fear of movement, graded activity, or exposure will be provided. When negative thoughts are recognized the adolescents are taught and trained on how to replace these thoughts, self-efficacy for target activities are increased by carefully selected activities witch allows the adolescent to succeed and by repeated feedback from the physiotherapists. Adequate coping strategies for restoring and sustaining activities are taught and trained. Parents are trained on how to support new behaviours.
* Applied skill acquisition The basic capabilities are put together in order to shape the more complex skills required when applying in target activities. Self- efficacy is reinforced by feedback from both the physiotherapists and parents.
* Generalisation This phase includes the generalisation of new, both physical and psychological skills to other, for the adolescent important, activities.
* Maintenance and relapse prevention This phase includes the identification of "risk situations", and recognition of how adolescents and parents can support positive behaviours further.

Patient follow-ups takes place immediately after completed intervention, after 6 months and after one year and two years after intervention in order to evaluate the long-term effect.

• Parents The treatment is based on earlier intervention program and includes; Information on pain and pain behaviours and parental impact on adolescent's pain behaviours. An individual intervention plan according to each teenager's problems is made. All parents will be trained on how to support new positive health behaviours.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents with pain and interference of daily activities due to pain, referred to paediatric physiotherapy in a primary health setting will be included.
* Participants must understand written and oral Swedish and have had persistent pain for more than 6 weeks or recurrent pain more than once a week for over three months.
* The adolescents´ parents will be included in a brief intervention.

Exclusion Criteria:

* Subjects with resent trauma, ongoing treatment for any psychiatric illness or cognitive problems will be excluded.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in Functional Disability Inventory | 6 months, one year and 2 years post treatment
  Functional Disability Inventory assesses children's self reported difficulties in physical and psychosocial functioning due to the child's physical health. FDI consists of 15 items describing limitations of activities during the past two weeks. Each item is scored on a 5-point (0-4) where a higher score indicates greater disability. The FDI has been reported to have a high validity and reliability and can be used for children and adolescents with recurrent and chronic pain.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Söderlund, Professor, Principal Investigator — Uppsala University
Locations (1):
- Samariterhemmet, Uppsala, Sweden